CLINICAL TRIAL: NCT00367926
Title: Effect of American Ginseng Root and Derived Polysaccharides on Postprandial Glycemia in Healthy Individuals
Brief Title: The Effect of American Ginseng Root and Its Components on Glycemia in Healthy Individuals
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Risk Factor Modification Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Ginseng Growers Association (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RFMC-0001-103; MOP- 62943
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2006-08-23 (Estimated); Status verified 2005-09

CONDITIONS: Hyperglycemia
Keywords: ginseng; polysaccharides; postprandial glycemia; area under the glucose curve; peak incremental glucose
MeSH Terms: conditions — Hyperglycemia | interventions — Polysaccharides

INTERVENTIONS:
Drug: American ginseng root / polysaccharides

SUMMARY:
To determine the effect of polysaccharides from American ginseng root on postprandial glycemia in healthy individuals.

DETAILED DESCRIPTION:
Glycemia-lowering effects of American ginseng root have been repeatedly observed in healthy individuals and in type 2 diabetes. It is unclear which components trigger these effects. Pre-clinical evidence suggests that, aside from ginseng saponins, ginseng polysaccharides may reduce glycemia. This assumption has not been investigated so far in humans.

We therefore undertook a double-blind randomized controlled clinical trial to determine the effect of American ginseng root polysaccharides, at escalating doses, on postprandial glycemia, in comparison to the American ginseng root and control in healthy individuals. We hypothesized that polysaccharides will reduce glycemia comparably to a dose of ginseng root that contains polysaccharides at an equivalent amount to the average polysaccharide dose. We therefore tested polysaccharide doses equivalent to 9, 12 and 15 g of rot, 12 go of ginseng root and a wheat bran control. Each subject received each treatment in random sequence, after a 12-hour overnight fast and 40 minutes prior to a 25-g oral glucose tolerance test. Capillary blood samples were collected at baseline, prior to glucose ingestion and at 15, 30, 45, 60, 90, 120 minutes after the start of glucose intake. Capillary blood glucose was measured.

ELIGIBILITY:
Inclusion Criteria:

* 16-65 years old
* normal renal and hepatic function
* fasting plasma glucose: 4-6 mmol/l
* clinically euthyroid
* normotensive

Exclusion Criteria:

* pregnant
* taking herbs, supplements or medication that affect glycemia
* major illnesses/ disease
* heavy alcohol use (> 3 drinks/ day)
* heavy smoking (> 10 cigarettes/ day)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 2005-06; Study Completion 2005-07

PRIMARY OUTCOMES:
incremental area under the postprandial glucose curve
incremental peak postprandial glucose

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, Ph.D., Principal Investigator — St. Michael's Hospital/ University of Toronto
Locations (1):
- Risk Factor Modification Centre, Toronto, Ontario, Canada